CLINICAL TRIAL: NCT02928315
Title: The Effect of Magnesium Therapy to Prevent Post-operative Atrial Fibrillation After Cardiac Surgery in Adults, Concerning the Perioperative Changes in Serum Electrolytes
Brief Title: The Effect of Magnesium Therapy to Prevent Post-operative Atrial Fibrillation After Cardiac Surgery in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00009907
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnesium (Active Comparator): Five ampules of 500 mg of magnesium sulfate will be dissolved in 100 ml of normal saline solution infused intravenously over 4 hours, once daily for 3 days starting when the patient is shifted to ICU.
  Interventions: Drug: Magnesium Sulfate
- control (Placebo Comparator): 100 ml of normal saline solution infused intravenously over 4 hours once daily , for 3 days
  Interventions: Other: control

INTERVENTIONS:
Drug: Magnesium Sulfate — The patients in the study group will receive 10 mmol of magnesium sulphate (2.47 gm). Five ampoules of 500 mg of magnesium sulphate will be dissolved in 100 ml of saline solution infused intravenously over 4 hours, once daily for 3 days starting when the patient is shifted to ICU.
  Arms: magnesium
Other: control — 100 ml of saline solution infused intravenously over 4 hours, once daily for 3 days starting when the patient is shifted to ICU.
  Arms: control

SUMMARY:
It is well known that magnesium sulfate has a membrane stabilizing effect , and broad spectrum anti arrhythmic properties. In this trial, the investigators study its prophylactic effect against atrial fibrillation in postoperative period of cardiac surgery.

DETAILED DESCRIPTION:
One of the most common postoperative complications after cardiac surgery is postoperative atrial fibrillation (AF). It is rarely fatal but it may cause subjective symptoms and result in thromboembolic complications, heart failure, renal insufficiency, and stroke which may prolong hospital stay.

The risk factors of AF include advanced age, transient atrial ischemia, arterial hypertension, dilated atria, male sex, pulmonary hypertension, previous atrial fibrillation and serum electrolyte disorders . On the other hand, there is evidence that cardiopulmonary bypass (CPB) time, duration of aortic cross clamping and the time of surgery, also the type of cardioplegia and the number of constructed grafts do not influence the incidence of AF.

There are only few studies that show the depletion of electrolytes and serum electrolyte concentration changes after cardiac surgery . The role of potassium in pathogenesis of cardiac arrhythmias is well recognized. Low serum potassium level is often found in association with hypomagnesemia and predisposes to atrial fibrillation. Extracellular magnesium is broadly implicated in neuronal control, neuromuscular transmission, and cardiovascular tone. It has been shown that magnesium suppresses arrhythmias after acute myocardial infarction, and there are studies confirming correlation between hypomagnesemia and postoperative atrial fibrillation . The underlying mechanism of these effects is not well understood but most probably involves magnesium interaction with calcium channels within myocytes membrane. Still the role of magnesium in the pathogenesis of AF is not clear yet.

Also, it is not clear if magnesium supplementation is useful for these patients, or it is useful only in hypomagnesemia patients. Hypophosphatemia and its consequences are less investigated in patients after cardiac surgery. Common complications after cardiac surgery are cardiac and respiratory failure, and they are also among the clinical manifestations of hypophosphatemia. Hypophosphatemia could be the cause of prolonged artificial lung ventilation and myocardial dysfunction; also, it may have influence on the incidence of arrhythmias. Anyway, there are no data confirming the arrhythmogenic effect of changes in serum phosphate level.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years.
* Left ventricular ejection fraction >0.3,
* Blood pressure is normal or less than 180/110.
* ASA ≤ III.
* Normal liver, pulmonary and renal function,
* No diabetes or other metabolism disorders,
* No pulmonary hypertension,
* No atrial fibrillation in the past, sinus rhythm on preoperative electrocardiogram.

Exclusion Criteria:

* history of AF,
* implanted pacemaker,
* postoperative myocardial infarction,
* use of left ventricular assist devices
* Renal failure or on hemodialysis

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | 3 post operative days
  the incidence of postoperative atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes